CLINICAL TRIAL: NCT05472012
Title: Performance of Masimo INVSENSOR00057 in Detecting Atrial Fibrillation (Afib)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ROBI0001
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Results first posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- INVSENSOR00057 (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00057 device.
  Interventions: Device: INVSENSOR00057

INTERVENTIONS:
Device: INVSENSOR00057 — Noninvasive wearable health monitoring device

SUMMARY:
This study is designed to validate the performance of Masimo INVSENSOR00057 in detecting atrial fibrillation. The noninvasive ECG measurements will be compared to results obtained from an FDA-cleared ECG monitor.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Subject is confirmed to have active atrial fibrillation at the time of enrollment.

Exclusion Criteria:

* Subject is confirmed to have concurrent active arrhythmias (e.g., PVCs, bradycardia, etc.) at the time of enrollment.
* Subject is allergic to adhesives or ECG gel.
* Subject whose skin is not intact in or at the vicinity of the device placement site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Site 1, Jackson, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00057
Started | 139
Completed | 139
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00057
Number analyzed (Participants) | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 119
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65
  Male | 74
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 134
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of INVSENSOR00057 Atrial Fibrillation (Afib) Detection Function
Description: Afib detection accuracy will be determined by analyzing the sensitivity of INVSENSOR00057 Afib detection function when compared to data collected using a FDA-cleared ECG monitor.
Time Frame: 1-5 hours
Population: A total of 23 subjects were excluded from the data analysis based on the protocol criteria. This included individuals whose reference or test ECG did not provide readable waveforms, as determined by medical personnel, and those who appeared to have atrial fibrillation (Afib) at enrollment but provided waveforms that were inconsistent with an Afib diagnosis.
Measure: Number; unit: % of true positive
Arm/Group | INVSENSOR00057
Number analyzed (Participants) | 116
% of true positive | 96.97

2. Primary Outcome: Specificity of INVSENSOR00057 Atrial Fibrillation (Afib) Detection Function
Description: Afib detection accuracy will be determined by analyzing the specificity of INVSENSOR00057 Afib detection function when compared to data collected using a FDA-cleared ECG monitor.
Time Frame: 1-5 hours
Population: as for outcome 1
Measure: Number; unit: % of true negative
Arm/Group | INVSENSOR00057
Number analyzed (Participants) | 116
% of true negative | 100

ADVERSE EVENTS:
Time Frame: 1-5 hours
Arm/Group | INVSENSOR00057
All-Cause Mortality (participants affected / at risk) | 0/139
Serious Adverse Events (participants affected / at risk) | 0/139
Other Adverse Events (participants affected / at risk) | 1/139
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INVSENSOR00057 (N=139)
Arm Cramp (Injury, poisoning and procedural complications) | 1 — The subject's arm experienced a cramp during the study, but the study continued once the cramp subsided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT05472012/Prot_SAP_000.pdf